CLINICAL TRIAL: NCT02016781
Title: A Multi-Center Biologic Assignment Trial Comparing Allogeneic Hematopoietic Cell Transplant to Hypomethylating Therapy or Best Supportive Care in Patients w/Intermediate-2 & High Risk Myelodysplastic Syndrome (BMTCTN1102)
Brief Title: Allo vs Hypomethylating/Best Supportive Care in MDS (BMTCTN1102)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN1102; 2U10HL069294-11 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2022-07-29 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: MDS
Keywords: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: Two arms will enroll and have data collected on them simultaneously.
Masking Description: No parties are masked in this trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transplant (Active Comparator): Reduced intensity conditioning allogeneic hematopoietic cell transplantation (RIC-alloHCT)
  Interventions: Procedure: Allogeneic Hematopoietic Cell Transplant
- Hypomethylating Therapy / Best Supportive Care (Active Comparator): The specific non-transplant treatment regimen will be at the discretion of the treating physician.
  Interventions: Procedure: Hypomethylating Therapy / Best Supportive Care

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Cell Transplant — Bone marrow or peripheral blood stem cell transplant.from a fully matched related (6/6) or unrelated (8/8) donor. The specific transplant treatment regimen will be at the discretion of the treating physician but is required to be reduced-intensity.
  Other Names: RIC alloHCT
  Arms: Transplant
Procedure: Hypomethylating Therapy / Best Supportive Care — The specific non-transplant treatment regimen will be at the discretion of the treating physician.
  Other Names: Non-transplant
  Arms: Hypomethylating Therapy / Best Supportive Care

SUMMARY:
This study is designed as a multicenter trial, with biological assignment to one of two study arms; Arm 1: Reduced intensity conditioning allogeneic hematopoietic cell transplantation (RIC-alloHCT), Arm 2: Non-Transplant Therapy/Best Supportive Care.

DETAILED DESCRIPTION:
Background: MDS is a clonal disorder of hematopoietic precursors and stem cells, which may evolve to a terminal phase resembling acute leukemia. A subject of clinical urgency for researchers, clinicians, patients, and health care underwriters such as Medicare, is the role of allogeneic hematopoietic cell transplantation (alloHCT) in the treatment of older patients with higher risk myelodysplastic syndromes (MDS). The use of reduced intensity conditioning (RIC) regimens has extended HCT to the care of older patients with acute myelogenous leukemia (AML) and lymphoma and a number of retrospective and phase II trials for patients with MDS now show the curative potential of RIC alloHCT in selected patients.

This protocol is designed to evaluate the relative benefits of RIC alloHCT compared to non-transplant therapies focusing on overall survival. This will be done by having patients biologically assigned to the alloHCT arm or the hypomethylating therapy/best supportive care arm and following them for survival at 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the following criteria will be eligible for entry into this study:

  1. Patients with de novo MDS who have, or have previously had, Intermediate-2 or High risk disease as determined by the International Prognostic Scoring System (IPSS). Current Intermediate-2 or High risk disease is NOT a requirement.
  2. Patients must have an acceptable MDS subtype:

     * Refractory cytopenia with unilineage dysplasia (RCUD) (includes refractory anemia (RA))
     * Refractory anemia with ringed sideroblasts (RARS)
     * Refractory anemia with excess blasts (RAEB-1)
     * Refractory anemia with excess blasts (RAEB-2)
     * Refractory cytopenia with multilineage dysplasia (RCMD)
     * Myelodysplastic syndrome with isolated del(5q) (5q-syndrome)
     * Myelodysplastic syndrome (MDS), unclassifiable
  3. Patients must have fewer than 20% marrow blasts within 60 days of consent.
  4. Patients may have received prior therapy for the treatment of MDS, including but not limited to: growth factor, transfusion support, immunomodulatory (IMID) therapy, DNA hypomethylating therapy, or cytotoxic chemotherapy prior to enrollment.
  5. Age 50.0-75.0 years.
  6. Karnofsky performance status > 70 or Eastern Cooperative Oncology Group (ECOG) ≤ 1.
  7. Patients are eligible if no formal unrelated donor search has been activated prior to date of consent. A formal unrelated donor search begins at the time at which samples are requested from potential National Marrow Donor Program (NMDP) donors. Patients who have started a sibling donor search or who have found a matched sibling donor are eligible.
  8. Patients and physicians must be willing to comply with treatment assignment:

     1. No intent to proceed with alloHCT using donor sources not specified in this protocol, including human leukocyte antigen (HLA)-mismatched related or unrelated donors (< 6/6 HLA related matched or < 8/8 HLA unrelated matched) or umbilical cord blood unit(s).
     2. No intent to use myeloablative conditioning regimens.
     3. Intent to proceed with RIC alloHCT if a matched sibling or matched unrelated donor is identified. There is no requirement as to the timing of the transplantation.
  9. Patients must be considered to be suitable RIC alloHCT candidates at the time of enrollment based on medical history, physical examination, and available laboratory tests. Specific testing for organ function is not required for eligibility but, if available, these tests should be used to judge eligibility.
  10. Signed informed consent

Exclusion Criteria:

* Patients with the following will be ineligible for registration onto this study:

  1. Therapy-related MDS (defined as the occurrence of MDS due to prior exposure to systemic chemotherapy and/or radiation for malignancy)
  2. Current or prior diagnosis of AML
  3. Chronic myelomonocytic leukemia or myelodysplastic/myeloproliferative neoplasm (unacceptable MDS subtypes); uncontrolled bacterial, viral or fungal infection (currently taking medication and with progression or no clinical improvement) at time of enrollment.
  4. Patients with prior malignancies, except treated non-melanoma skin cancer or treated cervical carcinoma in situ. Cancer treated with curative surgery without chemotherapy/radiation therapy > 5 years previously will be allowed. Cancer treated with curative surgery < 5 years previously will not be allowed unless approved by the Protocol Officer or one of the Protocol Chairs.
  5. Prior autologous or allogeneic HCT
  6. Human Immunodeficiency Virus (HIV) infection
  7. Patients of childbearing potential unwilling to use contraceptive techniques
  8. Patients with psychosocial conditions that would prevent study compliance

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research (CIBMTR), Medical College of Wisconsin
Locations (37):
- United States (37):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Florida College of Medicine, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland Medical Systems - Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute/Brigham & Women's, Boston, Massachusetts
  - Dana Farber Cancer Institute/Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute/BMT, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Jewish Hospital BMT Program, Cincinnati, Ohio
  - University Hospitals of Cleveland/ Case Western, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine/The Methodist Hospital, Houston, Texas
  - University of Texas/MD Anderson CRC, Houston, Texas
  - University of Utah Med School, Salt Lake City, Utah
  - Virginia Commonwealth University MCV Hospitals, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Saber W, Le Rademacher J, Sekeres M, Logan B, Lewis M, Mendizabal A, Leifer E, Appelbaum FR, Horowitz MM, Nakamura R, Cutler CS. Multicenter biologic assignment trial comparing reduced-intensity allogeneic hematopoietic cell transplant to hypomethylating therapy or best supportive care in patients aged 50 to 75 with intermediate-2 and high-risk myelodysplastic syndrome: Blood and Marrow Transplant Clinical Trials Network #1102 study rationale, design, and methods. Biol Blood Marrow Transplant. 2014 Oct;20(10):1566-72. doi: 10.1016/j.bbmt.2014.06.010. Epub 2014 Jun 24. PMID 24972249
- [Derived] Saber W, Bansal A, Li L, Scott BL, Sangaralingham LR, Thao V, Roth JA, Wright W, Steuten LMG, Pidala JA, Mishra A, Maziarz RT, Westervelt P, McGuirk JP, Cutler C, Nakamura R, Ramsey SD. Cost-Effectiveness of Reduced-Intensity Allogeneic Hematopoietic Cell Transplantation for Older Patients With High-Risk Myelodysplastic Syndrome: Analysis of BMT CTN 1102. JCO Oncol Pract. 2024 Apr;20(4):572-580. doi: 10.1200/OP.23.00413. Epub 2024 Jan 23. PMID 38261970
- [Derived] Versluis J, Saber W, Tsai HK, Gibson CJ, Dillon LW, Mishra A, McGuirk J, Maziarz RT, Westervelt P, Hegde P, Mukherjee D, Martens MJ, Logan B, Horowitz M, Hourigan CS, Nakamura R, Cutler C, Lindsley RC; Blood and Marrow Transplant Clinical Trials Network. Allogeneic Hematopoietic Cell Transplantation Improves Outcome in Myelodysplastic Syndrome Across High-Risk Genetic Subgroups: Genetic Analysis of the Blood and Marrow Transplant Clinical Trials Network 1102 Study. J Clin Oncol. 2023 Oct 1;41(28):4497-4510. doi: 10.1200/JCO.23.00866. Epub 2023 Aug 22. PMID 37607457
- [Derived] Cusatis R, Martens MJ, Nakamura R, Cutler CS, Saber W, Lee SJ, Logan BR, Shaw BE, Gregory A, D'Souza A, Hamilton BK, Horowitz MM, Flynn KE. Health-related quality of life in reduced-intensity hematopoietic cell transplantation based on donor availability in patients aged 50-75 with advanced myelodysplastic syndrome: BMT CTN 1102. Am J Hematol. 2023 Feb;98(2):229-250. doi: 10.1002/ajh.26768. Epub 2022 Nov 21. PMID 36251401
- [Derived] Nakamura R, Saber W, Martens MJ, Ramirez A, Scott B, Oran B, Leifer E, Tamari R, Mishra A, Maziarz RT, McGuirk J, Westervelt P, Vasu S, Patnaik M, Kamble R, Forman SJ, Sekeres MA, Appelbaum F, Mendizabal A, Logan B, Horowitz M, Cutler C. Biologic Assignment Trial of Reduced-Intensity Hematopoietic Cell Transplantation Based on Donor Availability in Patients 50-75 Years of Age With Advanced Myelodysplastic Syndrome. J Clin Oncol. 2021 Oct 20;39(30):3328-3339. doi: 10.1200/JCO.20.03380. Epub 2021 Jun 9. PMID 34106753
- See also: National Marrow Donor Program — http://bethematch.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 34 centers between December 2013 and November 2018. The study opened to accrual on December 16, 2013 with 36 centers activated for enrollment. The study closed to accrual on November 9, 2018 and study completed on October 5, 2021.
Pre-assignment Details: Participants whose donors were found during the search were assigned to HCT arm. Participants whose donors were not found by the end of the search were assigned to Non-HCT arm.
Groups:
- HCT Arm: Reduced intensity conditioning allogeneic hematopoietic cell transplantation (RIC-alloHCT)
  All subjects are initially assigned to the non-transplant arm. Subjects are re-assigned to the transplant arm should a suitable donor be identified within 90 days of informed consent.
  Bone marrow or peripheral blood stem cell transplant from a fully matched related (6/6) or unrelated (8/8) donor. Donors must meet institutional selection criteria, and there is no age restriction for sibling donors. The specific transplant treatment regimen will be at the discretion of the treating physician but is required to be reduced-intensity.
  The following limits on conditioning dose intensity delineate myeloablative regimens:
  1. TBI doses of ≥ 500 (unfractionated) cGy and ≥ 800 cGy (fractionated)
     All supportive care will be given in keeping with the BMT CTN Manual of Procedures (MOP) and local institutional guidelines. All patients will receive prophylaxis against bacterial, fungal, and viral infections during the post-HCT period according to institutional standards.
  2. Busulfan dose ≥ 9.5 mg/kg
  3. Melphalan ≥ 150 mg/m2
- Non-HCT Arm: Non-Transplant Therapy/Best Supportive Care The specific non-transplant treatment regimen will be at the discretion of the treating physician.
  Hypomethylating therapy is the accepted standard therapy of treatment naïve patients with Int-2/High Risk MDS not undergoing transplantation. Azacytidine: 75 mg/m2 by subcutaneous injection or IV for 7 days; 28 day cycles. Or Decitabine: 20 mg/m2 IV daily for 5 days; 28 day cycles.
  All supportive care will be given in keeping with local institutional guidelines.
Period: Interim Look for Primary Analysis
Arm/Group | HCT Arm | Non-HCT Arm
Started (Interim look uses data cutoff as of February 18, 2020) | 260 | 124
Completed (Patients completed 3 years of follow up or died.) | 187 | 100
Not Completed | 73 | 24
Not completed — Alive and on study | 71 | 23
Not completed — Withdrawal by Subject | 2 | 1
Period: Final Database Lock
Arm/Group | HCT Arm | Non-HCT Arm
Started (Final database lock was on May 24, 2022. One patient was categorized in the non-HCT arm at interim analysis data look. The site corrected data to assign this patient to HCT arm after interim analysis data cutoff date and confirmed that the patient did receive transplant. Patients missing visits or data was unable to be obtained are categorized as not completing the study due to missing data.) | 261 | 123
Completed | 248 | 115
Not Completed | 13 | 8
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 11 | 4
Not completed — Missing data | 0 | 3

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes intent to treat (ITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | HCT Arm | Non-HCT Arm | Total
Number analyzed (Participants) | 260 | 124 | 384
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 105 | 44 | 149
  >=65 years | 155 | 80 | 235
Age, Continuous [Mean (Standard Deviation); unit: year] | 65.6 (5.6) | 66.0 (5.9) | 65.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 48 | 143
  Male | 165 | 76 | 241
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 233 | 108 | 341
  Unknown or Not Reported | 16 | 7 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 8 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 234 | 105 | 339
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 7 | 18
Karnofsky Performance Score (KPS) [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead Population: Either KPS or ECOG were collected from each participant at enrollment, not both.
  Participants
    number analyzed (Participants) | 180 | 84 | 264
    >=90 | 99 | 35 | 134
    <90 | 81 | 49 | 130
ECOG Performance Score [Count of Participants; unit: Participants] — It measures how the disease impacts a patient's daily living abilities a scale of 0-5.
  0: Fully active, able to carry on all pre-disease activities without restriction; 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about >50% of waking hours; 3: Capable of only limited selfcare, confined to bed or chair > 50% of waking hours; 4: Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair; 5: Dead. Population: Either KPS or ECOG were collected from each participant at enrollment, not both.
  Participants
    number analyzed (Participants) | 80 | 40 | 120
    0 | 24 | 16 | 40
    > 0 | 56 | 24 | 80
MDS Subtype [Count of Participants; unit: Participants]
  Refractory cytopenia with unilineage dysplasia (RCUD) | 5 | 1 | 6
  Refractory anemia with ringed sideroblasts (RARS) | 5 | 2 | 7
  Refractory anemia with excess blasts (RAEB-1) | 61 | 31 | 92
  Refractory anemia with excess blasts (RAEB-2) | 132 | 63 | 195
  Refractory cytopenia with multilineage dysplasia (RCMD) | 36 | 14 | 50
  Myelodysplastic syndrome with isolated del(5q) (5q-syndrome) | 6 | 7 | 13
  Myelodysplastic syndrome (MDS), unclassifiable | 15 | 6 | 21
MDS Duration from Diagnosis to Enrollment (months) [Mean (Standard Deviation); unit: months] | 8.4 (21.6) | 11.0 (27.1) | 9.2 (23.5)
Identified Donor Type (HCT Arm only) [Count of Participants; unit: Participants] — Population: Donor type is only available for HCT arm.
  Participants
    number analyzed (Participants) | 260 | 0 | 260
    HLA Matched Related | 80 | 0 | 80
    HLA Matched Unrelated | 180 | 0 | 180
Donor Gender (HCT Arm only) [Count of Participants; unit: Participants] — Population: Donor gender is only available for HCT arm.
  Participants
    number analyzed (Participants) | 260 | 0 | 260
    Female | 73 | 0 | 73
    Male | 130 | 0 | 130
    Missing | 57 | 0 | 57
HCT-CI (HCT Arm only) [Count of Participants; unit: Participants] — The HCT-CI was developed to identify comorbidities relevant to transplant and act as a tool for risk assessment and before allogeneic hematopoietic stem cell transplantation. Patients with no comorbidities are assigned a score of zero. Arrhythmia, cardiac, bowel, diabetes, cerebrovascular, psychological, mild chronic hepatitis, obesity, infection are assigned a score of 1. Rheumatoid arthritis, peptic ulcer, renal moderate/severe, pulmonary moderate, are assigned a score of 2. Solid tumor, heart valve disease, pulmonary sever, hepatic moderate/severe are assigned a score of 3. Population: HCT-CI is only available for HCT arm.
  Participants
    number analyzed (Participants) | 260 | 0 | 260
    0 | 41 | 0 | 41
    1 | 31 | 0 | 31
    2 | 35 | 0 | 35
    3 | 98 | 0 | 98
    Missing | 55 | 0 | 55
Highest IPSS Score [Count of Participants; unit: Participants] — The International Prostate Symptom Score (IPSS) determines the prognosis of patients with MDS. It guides clinicians and patients in determining the optimal risk-adapted treatment strategy. Covariates for prognostic discrimination include percentage of bone marrow blasts, Karyotype, and number of cytopenias at the time of initial diagnosis, which distinguish four prognostic categories of low-risk (IPSS: 0), intermediate-1 (IPSS: 0.5-1), intermediate-2 (IPSS: 1.5-2), and high-risk disease (IPSS: >=2.5).
  Participants
    Intermediate-2 (1.5-2.0) | 173 | 81 | 254
    High Risk (>=2.5) | 87 | 43 | 130
Highest IPSS-R Score [Count of Participants; unit: Participants] — Revised International Prognostic Scoring System (IPSS-R) for MDS further refines the prognostic value of IPSS. IPSS-R utilizes the IPSS platform, with the addition of seven chromosomal abnormalities, further discrimination of the percentage of bone marrow blasts, and incorporation of the severity of each cytopenia to create five cytogenetic risk groups: Very low (<=1.5), Low (>1.5-3.0), Intermediate (>3-4.5), High (>4.5-6), Very High (>6).
  Participants
    Very Low | 4 | 0 | 4
    Low | 2 | 0 | 2
    Intermediate | 79 | 34 | 113
    High | 82 | 51 | 133
    Very High | 93 | 39 | 132
Response to Hypomethylating Therapy [Count of Participants; unit: Participants] — Response is defined as achieving complete response, partial response, or hematologic improvement, or no response.
  Participants
    Complete Response | 10 | 7 | 17
    Partial Response | 46 | 23 | 69
    No Response | 79 | 42 | 121
    Never had therapy | 88 | 33 | 121
    Unknown | 37 | 19 | 56
Cytogenetics Tested [Count of Participants; unit: Participants]
  Yes | 241 | 112 | 353
  No | 12 | 8 | 20
  Unknown or Missing | 7 | 4 | 11
Results of Cytogenetics Test [Count of Participants; unit: Participants] — Population: Results of cytogenetics test is only available for participants who had cytogenetics tested.
  Participants
    number analyzed (Participants) | 241 | 112 | 353
    Abnormalities Identified | 151 | 81 | 232
    No Evaluable Metaphases | 4 | 0 | 4
    No Abnormalities | 84 | 31 | 115
    Missing | 2 | 0 | 2
Number of Distinct Cytogenetic Abnormalities [Count of Participants; unit: Participants] — Population: Number of distinct cytogenetic abnormalities is only available for participants who had a abnormalities cytogenetics test result.
  Participants
    number analyzed (Participants) | 151 | 81 | 232
    1 | 43 | 28 | 71
    2 | 31 | 19 | 50
    3 | 20 | 14 | 34
    >=4 | 52 | 20 | 72
    Missing | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Survival (OS)
Description: The primary endpoint for this study is overall survival (OS) at three years post-consent. Death from any cause will be considered an event for this endpoint. Surviving participants are censored at the time of last follow-up. Three year OS estimates are adjusted for age, race/ethnicity, performance status, IPSS score, duration of disease, and response to prior hypomethylating therapy. The results posted are from the February 2020 interim analysis per protocol study design. Two interim analyses for efficacy were performed previously in January and November 2019 and presented to the Data and Safety Monitoring Board (DSMB). Results at the second analysis was crossing the efficacy boundary. Subsequently, the DSMB approved early release of study data as of February 2020.
Time Frame: 3 years
Population: The enrolled participants are included in the analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 260 | 124
percentage of participants | 47.9 [41.3 to 54.1] | 26.6 [18.4 to 35.6]
Statistical Analysis 1: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the rates of three-year OS are the same for both treatments. The results posted are from the interim analysis per protocol study design; Test type: Superiority; p = 0.0001, Wald test — Statistical significance was determined using a pre-specified threshold of 0.05; Wald test of difference in adjusted OS estimates
Statistical Analysis 2: Comparison: HCT Arm vs Non-HCT Arm; This subgroup analysis investigated the differential impact of response to hypomethylating therapy (No Response to Hypomethylation vs. Any Response or Hematologic Improvement to Hypomethylation vs. No Prior Hypomethylation) on the treatment effect for OS at three years post-consent for the HCT arm vs. the non-HCT arm. The analysis was conducted using pseudo-value regression models via an interaction term between the factor and the treatment group with a logit link function; Test type: Superiority; p = 0.3345, pseudo-value regression models — Statistical significance was determined using a pre-specified threshold of 0.05; Overall Wald test of interaction terms between response to hypomethylating therapy and treatment assignment in regression model
Statistical Analysis 3: Comparison: HCT Arm vs Non-HCT Arm; This subgroup analysis investigated the differential impact of patient age (< vs. >= 65) on the treatment effect for OS at three years post-consent for the HCT arm vs. the non-HCT arm. The analysis was conducted using pseudo-value regression models via an interaction term between the factor and the treatment group with a logit link function; Test type: Superiority; p = 0.7328, pseudo-value regression models — Statistical significance was determined using a pre-specified threshold of 0.05; Overall Wald test of interaction terms between patient age and treatment assignment in regression model
Statistical Analysis 4: Comparison: HCT Arm vs Non-HCT Arm; This subgroup analysis investigated the differential impact of disease duration (less than vs. 3 months or more) on the treatment effect for OS at three years post-consent for the HCT arm vs. the non-HCT arm. The analysis was conducted using pseudo-value regression models via an interaction term between the factor and the treatment group with a logit link function; Test type: Superiority; p = 0.6261, pseudo-value regression models — Statistical significance was determined using a pre-specified threshold of 0.05; Overall Wald test of interaction terms between disease duration and treatment assignment in regression model
Statistical Analysis 5: Comparison: HCT Arm vs Non-HCT Arm; This subgroup analysis investigated the differential impact of IPSS score (Intermediate-2 vs. High) on the treatment effect for OS at three years post-consent for the HCT arm vs. the non-HCT arm. The analysis was conducted using pseudo-value regression models via an interaction term between the factor and the treatment group with a logit link function; Test type: Superiority; p = 0.4134, pseudo-value regression models — Statistical significance was determined using a pre-specified threshold of 0.05; Overall Wald test of interaction terms between IPSS score and treatment assignment in regression model
Statistical Analysis 6: Comparison: HCT Arm vs Non-HCT Arm; Statistical Analysis 6: This subgroup analysis investigated the differential impact of IPSS-R score (Very Low, Low, or Intermediate vs. High vs. Very High) on the treatment effect for OS at three years post-consent for the HCT arm vs. the non-HCT arm. The analysis was conducted using pseudo-value regression models via an interaction term between the factor and the treatment group with a logit link function; Test type: Superiority; p = 0.3147, pseudo-value regression models — Statistical significance was determined using a pre-specified threshold of 0.05; Overall Wald test of interaction terms between IPSS-R score and treatment assignment in regression model

2. Secondary Outcome: Percentage of Participants With Leukemia-free Survival (LFS)
Description: LFS is defined as the time from the date of patient consent to the date of progression to AML or death from any cause, whichever comes first. Progression to AML is defined as > 20% leukemic blasts in bone marrow or in the peripheral blood. Death from any cause or transformation of MDS to AML are considered events for this endpoint. Participants without either event are censored at the time of last follow-up. Three year leukemia-free survival probability estimates are adjusted for age, race/ethnicity, performance status, IPSS score, duration of disease, and response to prior hypomethylating therapy.
Time Frame: 3 years
Population: The enrolled participants are included in the analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 260 | 124
percentage of participants | 35.8 [29.8 to 41.8] | 20.6 [13.3 to 29.1]
Statistical Analysis 1: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the rates of three-year LFS are the same for both treatments; Test type: Superiority; p = 0.0030, Wald test — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: HCT Arm vs Non-HCT Arm; This subgroup analysis investigated the differential impact of response to hypomethylating therapy on the treatment effect for LFS at three years post-consent for the HCT arm vs. the non-HCT arm. The analysis was conducted using pseudo-value regression models via an interaction term between the factor and the treatment group with a logit link function; Test type: Superiority; p = 0.9908, pseudo-value regression models — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 3: Comparison: HCT Arm vs Non-HCT Arm; This subgroup analysis investigated the differential impact of patient age (< or >= 65) on the treatment effect for LFS at three years post-consent for the HCT arm vs. the non-HCT arm. The analysis was conducted using pseudo-value regression models via an interaction term between the factor and the treatment group with a logit link function; Test type: Superiority; p = 0.8981, pseudo-value regression models — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 4: Comparison: HCT Arm vs Non-HCT Arm; This subgroup analysis investigated the differential impact of disease duration (less than vs. 3 months or more) on the treatment effect for LFS at three years post-consent for the HCT arm vs. the non-HCT arm. The analysis was conducted using pseudo-value regression models via an interaction term between the factor and the treatment group with a logit link function; Test type: Superiority; p = 0.1465, pseudo-value regression models — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 5: Comparison: HCT Arm vs Non-HCT Arm; This subgroup analysis investigated the differential impact of IPSS score (Intermediate-2 vs. High) on the treatment effect for LFS at three years post-consent for the HCT arm vs. the non-HCT arm. The analysis was conducted using pseudo-value regression models via an interaction term between the factor and the treatment group with a logit link function; Test type: Superiority — Statistical significance was determined using a pre-specified threshold of 0.05; p = 0.4991, pseudo-value regression models
Statistical Analysis 6: Comparison: HCT Arm vs Non-HCT Arm; This subgroup analysis investigated the differential impact of IPSS-R score on the treatment effect for LFS at three years post-consent for the HCT arm vs. the non-HCT arm. The analysis was conducted using pseudo-value regression models via an interaction term between the factor and the treatment group with a logit link function; Test type: Superiority; p = 0.4953, pseudo-value regression models — Statistical significance was determined using a pre-specified threshold of 0.05

3. Secondary Outcome: Quality of Life (QOL) - Functional Assessment of Cancer Therapy-General (FACT-G)
Description: QOL will be compared between the 2 arms using the FACT-G instrument. FACT-G evaluates the health-related quality of life (HQL) of patients receiving treatment for cancer. FACT-G consists of four subscales developed and normed in cancer patients: Physical Well-being, Social/Family Well-being, Emotional Well-being, and Functional Well-being. The FACT-G score ranges 0-108. Each subscale is positively scored, with higher scores indicating better functioning. The self-reported questionnaire will be completed at enrollment and at 6, 12, 18, 24, and 36 months from consent. Results shown are FACT-G total scores.
Time Frame: 3 years
Population: The enrolled participants are included in the analyses. Only English and Spanish speaking patients were eligible to participate in the QOL component of this trial.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 260 | 124
score on a scale
  Enrollment: number analyzed (Participants) | 203 | 86
  Enrollment | 81.5 (1.1) | 79.3 (1.9)
  6 Months: number analyzed (Participants) | 173 | 70
  6 Months | 81.4 (1.1) | 78.6 (2.0)
  12 Months: number analyzed (Participants) | 134 | 46
  12 Months | 84.0 (1.2) | 80.8 (2.2)
  18 Months: number analyzed (Participants) | 101 | 36
  18 Months | 87.7 (1.5) | 83.8 (2.8)
  24 Months: number analyzed (Participants) | 79 | 24
  24 Months | 89.0 (1.6) | 87.0 (3.4)
  36 Months: number analyzed (Participants) | 58 | 11
  36 Months | 90.3 (2.0) | 79.7 (5.9)
Statistical Analysis 1: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the FACT-G scores are the same at Enrollment for both treatments; Test type: Superiority; p = 0.2777, t-test, 2 sided — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in FACT-G scores from enrollment are the same at 6 Months for both treatments; Test type: Superiority; p = 0.2250, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; Changes in scores from enrollment were compared between arms using ANOVA models with treatment arm as main effect and enrollment score as a covariate
Statistical Analysis 3: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in FACT-G scores from enrollment are the same at 12 Months for both treatments; Test type: Superiority; p = 0.1048, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in FACT-G scores from enrollment are the same at 18 Months for both treatments; Test type: Superiority; p = 0.0888, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in FACT-G scores from enrollment are the same at 24 Months for both treatments; Test type: Superiority; p = 0.5844, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in FACT-G scores from enrollment are the same at 36 Months for both treatments; Test type: Superiority; p = 0.0344, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]

4. Secondary Outcome: Quality of Life (QOL) - Medical Outcomes Study Short Form (MOS SF-36)
Description: SF36 is being used in this protocol as a generic measure of quality of life (QOL). The self-reported questionnaires are completed at enrollment and at 6, 12, 18, 24, and 36 months from consent. The MOS SF-36 instrument is a general assessment of health QOL with eight components: Physical Functioning, Role Physical, Pain Index, General Health Perceptions, Vitality, Social Functioning, Role Emotional, and Mental Health Index. The sub scores for each of the eight components were computed based on the raw categorical values from the survey and range 0-100 with higher scores indicating better outcomes for each domain. Then overall Physical Component Summary (PCS) and Mental Component Summary (MCS) are computed using standardized algorithm for SF36. MCS and PCS scores range 0-100 with higher score indicating positive outcome. To facilitate comparison of the results with published norms, PCS and MCS are used as the outcome measures in summarizing the SF-36 data.
Time Frame: 3 years
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 260 | 124
score on a scale
  PCS at Enrollment: number analyzed (Participants) | 198 | 85
  PCS at Enrollment | 38.8 (0.8) | 37.9 (1.2)
  PCS at 6 Months: number analyzed (Participants) | 167 | 71
  PCS at 6 Months | 38.1 (0.7) | 37.8 (1.2)
  PCS at 12 Months: number analyzed (Participants) | 132 | 44
  PCS at 12 Months | 39.9 (0.8) | 37.7 (1.8)
  PCS at 18 Months: number analyzed (Participants) | 101 | 36
  PCS at 18 Months | 42.1 (0.9) | 40.5 (1.6)
  PCS at 24 Months: number analyzed (Participants) | 78 | 24
  PCS at 24 Months | 43.2 (1.1) | 41.2 (2.3)
  PCS at 36 Months: number analyzed (Participants) | 59 | 11
  PCS at 36 Months | 44.0 (1.3) | 39.3 (3.9)
  MCS at Enrollment: number analyzed (Participants) | 198 | 85
  MCS at Enrollment | 49.9 (0.8) | 50.7 (1.0)
  MCS at 6 Months: number analyzed (Participants) | 167 | 71
  MCS at 6 Months | 50.1 (0.8) | 50.7 (1.4)
  MCS at 12 Months: number analyzed (Participants) | 132 | 44
  MCS at 12 Months | 52.6 (0.8) | 53.4 (1.2)
  MCS at 18 Months: number analyzed (Participants) | 101 | 36
  MCS at 18 Months | 54.4 (0.9) | 52.0 (1.7)
  MCS at 24 Months: number analyzed (Participants) | 78 | 24
  MCS at 24 Months | 54.4 (0.9) | 53.2 (1.4)
  MCS at 36 Months: number analyzed (Participants) | 59 | 11
  MCS at 36 Months | 54.0 (1.1) | 53.6 (4.4)
Statistical Analysis 1: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the MOS SF-36 PCS scores are the same at Enrollment for both treatments; Test type: Superiority; p = 0.5583, t-test, 2 sided — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in MOS SF-36 PCS scores from enrollment are the same at 6 Months for both treatments; Test type: Superiority; p = 0.6690, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in MOS SF-36 PCS scores from enrollment are the same at 12 Months for both treatments; Test type: Superiority; p = 0.2089, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in MOS SF-36 PCS scores from enrollment are the same at 18 Months for both treatments; Test type: Superiority; p = 0.4343, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in MOS SF-36 PCS scores from enrollment are the same at 24 Months for both treatments; Test type: Superiority; p = 0.5942, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in MOS SF-36 PCS scores from enrollment are the same at 36 Months for both treatments; Test type: Superiority; p = 0.1615, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 7: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the MOS SF-36 MCS scores are the same at Enrollment for both treatments; Test type: Superiority; p = 0.5659, t-test, 2 sided — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 8: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in MOS SF-36 MCS scores from enrollment are the same at 6 Months for both treatments; Test type: Superiority; p = 0.8555, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 9: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in MOS SF-36 MCS scores from enrollment are the same at 12 Months for both treatments; Test type: Superiority; p = 0.8995, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 10: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in MOS SF-36 MCS scores from enrollment are the same at 18 Months for both treatments; Test type: Superiority; p = 0.0105, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 11: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in MOS SF-36 MCS scores from enrollment are the same at 24 Months for both treatments; Test type: Superiority; p = 0.2596, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 12: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in MOS SF-36 MCS scores from enrollment are the same at 36 Months for both treatments; Test type: Superiority; p = 0.5022, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]

5. Secondary Outcome: Quality of Life (QOL) - EQ-5D
Description: QOL will be compared between the 2 arms using the EQ-5D survey. The EQ-5D contains a five-item survey with three response levels per item measuring mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D takes approximately 1 minute to complete (Agency for Healthcare Research and Quality, 2005). The EQ-5D score ranges -0.224 to 1. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. The self-reported questionnaire will be completed at enrollment and at 6, 12, 18, 24, and 36 months from consent.
Time Frame: 3 years
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 260 | 124
score on a scale
  Enrollment: number analyzed (Participants) | 202 | 86
  Enrollment | 0.800 (0.010) | 0.823 (0.015)
  6 Months: number analyzed (Participants) | 169 | 72
  6 Months | 0.779 (0.013) | 0.792 (0.020)
  12 Months: number analyzed (Participants) | 133 | 47
  12 Months | 0.792 (0.014) | 0.772 (0.028)
  18 Months: number analyzed (Participants) | 102 | 37
  18 Months | 0.826 (0.016) | 0.812 (0.025)
  24 Months: number analyzed (Participants) | 79 | 24
  24 Months | 0.845 (0.016) | 0.858 (0.034)
  36 Months: number analyzed (Participants) | 59 | 11
  36 Months | 0.835 (0.024) | 0.789 (0.061)
Statistical Analysis 1: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the EQ-5D scores are the same at Enrollment for both treatments; Test type: Superiority; p = 0.1768, t-test, 2 sided — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in EQ-5D scores from enrollment are the same at 6 Months for both treatments; Test type: Superiority; p = 0.8318, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in EQ-5D scores from enrollment are the same at 12 Months for both treatments; Test type: Superiority; p = 0.4752, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in EQ-5D scores from enrollment are the same at 18 Months for both treatments; Test type: Superiority; p = 0.5671, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in EQ-5D scores from enrollment are the same at 24 Months for both treatments; Test type: Superiority; p = 0.3009, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the changes in EQ-5D scores from enrollment are the same at 36 Months for both treatments; Test type: Superiority; p = 0.3403, ANOVA — Statistical significance was determined using a pre-specified threshold of 0.05; [statistical method as in outcome 3, analysis 2]

6. Secondary Outcome: Percentage of Participants With Overall Survival (OS) in As-treated Population
Description: Time to event outcomes will be analyzed from the time of consent. Death from any cause will be considered an event for this endpoint. Surviving participants are censored at the time of last follow-up. Three-year OS estimates are adjusted for age, race/ethnicity, performance status, IPSS score, duration of disease, and response to prior hypomethylating therapy.
Time Frame: 3 years
Population: The treated participants are included in the analyses. This secondary analysis includes only treated participants who were compliant with their biologic assignment during the first six months following final assignment and excludes participants from the analysis if they died or dropped out before 90 days without a donor identified.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 216 | 85
percentage of participants | 49.4 [42.6 to 55.9] | 17.4 [9.4 to 27.5]
Statistical Analysis 1: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the rates of three-year OS are the same for both treatments in treated population; Test type: Superiority; p < 0.0001, Wald test — Statistical significance was determined using a pre-specified threshold of 0.05

7. Secondary Outcome: Percentage of Participants With Leukemia-free Survival (LFS) in As-treated Population
Description: as for outcome 2
Time Frame: 3 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 216 | 85
percentage of participants | 39.5 [32.9 to 46.1] | 11.2 [4.6 to 21.3]
Statistical Analysis 1: Comparison: HCT Arm vs Non-HCT Arm; The null hypothesis is that the rates of three-year LFS are the same for both treatments in treated population; Test type: Superiority; p < 0.0001, Wald test — Statistical significance was determined using a pre-specified threshold of 0.05

8. Secondary Outcome: Percentage of Participants on HCT Arm With Overall Survival (OS)
Description: The time to event outcomes is evaluated from the time of transplant. Death from any cause will be considered an event for this endpoint. Surviving participants are censored at the time of last follow-up. OS estimates are adjusted for age, race/ethnicity, performance status, IPSS score, duration of disease, and response to prior hypomethylating therapy.
Time Frame: 27 months post-transplant
Population: The enrolled participants in the HCT arm who received HCT from their assigned donor.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 216 | 0
percentage of participants | 55.7 [48.4 to 62.4] |

9. Secondary Outcome: Percentage of Participants on HCT Arm With Disease Relapse
Description: Outcome Measure Description: The time to event outcomes is evaluated from the time of transplant. Disease relapse is defined as: Satisfying criteria for evolution into acute leukemia; or reappearance of pre-transplant morphologic abnormalities, detected in bone marrow specimens; or reappearance of pre-transplant cytogenetic abnormality in at least one metaphase on each of two separate consecutive examinations at least one month apart, regardless of the number of metaphases analyzed; or institution of any therapy to treat relapsed disease (institution of any therapy not meant for maintenance or prevention), including withdrawal of immunosuppressive therapy or DLI. Relapse estimates are adjusted for age, race/ethnicity, performance status, IPSS score, duration of disease, and response to prior hypomethylating therapy.
Time Frame: 27 months post-transplant
Population: The enrolled participants in the HCT arm who received HCT from their assigned donor.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 216 | 0
percentage of participants | 29.6 [23.5 to 35.9] |

10. Secondary Outcome: Percentage of Participants on HCT Arm With Disease-free Survival (DFS)
Description: The time to event outcomes is evaluated from the time of transplant. Death or disease relapse/progression will be considered as events for this endpoint. Surviving participants are censored at the time of last follow-up. DFS estimates are adjusted for age, race/ethnicity, performance status, IPSS score, duration of disease, and response to prior hypomethylating therapy.
Time Frame: 27 months post-transplant
Population: The enrolled participants in the HCT arm who received HCT from their assigned donor.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 216 | 0
percentage of participants | 49.7 [42.6 to 56.5] |

11. Secondary Outcome: Percentage of Participants on HCT Arm With Treatment-related Mortality
Description: The time to event outcomes is evaluated from the time of transplant. The events are deaths prior to disease relapse. TRM estimates are adjusted for age, race/ethnicity, performance status, IPSS score, duration of disease, and response to prior hypomethylating therapy.
Time Frame: 27 months post-transplant
Population: The enrolled participants in the HCT arm who received HCT from their assigned donor.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 216 | 0
percentage of participants | 20.6 [15.3 to 26.5] |

12. Secondary Outcome: Percentage of Participants on HCT Arm With Grade II-IV Acute GVHD (aGVHD)
Description: Grade II-IV aGVHD is the event. aGVHD will be graded according to the BMT CTN Manual of Procedures (MOP). Staging for skin: Stage 1. <25% rash; 2. 25-50%; 3. >50%; 4. generalized erythroderma with bullae. Staging for GI: Stage 1. Diarrhea>500ml/d or persistent nausea; 2. >1000ml/d; 3. >1500ml/d; 4. Large volume diarrhea and severe abdominal pain +- ileus. Staging for Liver: Stage 1. bilirubin 2-3mg/dl; 2. bilirubin 3-6 mg/dl; 3. bilirubin 6-15 mg/dl; 4. bilirubin>15mg/dl. aGVHD grading is performed by the consensus conference criteria (Przepiorka et al. 1995). Grade I aGVHD is defined as Skin stage of 1-2 and stage 0 for both GI and liver organs. Grade II is stage 3 of skin, or stage 1 of GI, or stage 1 of liver. Grade III is stage 2-4 for GI, or stage 2-3 of liver. Grade IV is stage 4 of skin, or stage 4 of liver.
Time Frame: 27 months post-transplant
Population: Enrolled participants in the HCT arm who received HCT from their assigned donor and who had Grade II-IV Acute GVHD data from CIBMTR are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 201 | 0
percentage of participants | 43.1 [36.1 to 49.9] |

13. Secondary Outcome: Percentage of Participants on HCT Arm With Grade III-IV Acute GVHD
Description: The time to event outcomes is evaluated from the time of transplant. Grade III-IV Acute GVHD will be considered as events for this endpoint.
Time Frame: 27 months post-transplant
Population: Enrolled participants in the HCT arm who received HCT from their assigned donor and who had Grade III-IV Acute GVHD data from CIBMTR are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 201 | 0
percentage of participants | 17.1 [12.2 to 22.7] |

14. Secondary Outcome: Percentage of Participants on HCT Arm With Chronic GVHD
Description: The time to event outcomes is evaluated from the time of transplant. Chronic GVHD will be considered as events for this endpoint. Data will be collected and reviewed according to the recommendations of the NIH Consensus Criteria. Eight organs will be scored on a 0-3 scale to reflect degree of chronic GVHD involvement. Liver and pulmonary function test results and use of systemic therapy for treatment of chronic GVHD will also be recorded. This secondary endpoint of chronic GVHD will include mild, moderate and severe chronic GVHD based on NIH Consensus Criteria.
Time Frame: 27 months post-transplant
Population: Enrolled participants in the HCT arm who received HCT from their assigned donor and who had Chronic GVHD data from CIBMTR are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCT Arm | Non-HCT Arm
Number analyzed (Participants) | 202 | 0
percentage of participants | 55.5 [47.8 to 62.5] |

ADVERSE EVENTS:
Time Frame: Adverse event reporting and monitoring were conducted throughout the study, up to 3 years.
Description: Per Protocol 4.4.5. AE Reporting, no other therapy is mandated in this study, AE associated with transplantation or non-transplantation will not be collected nor reported for this protocol. Only AE related to the study consent process, collection of the optional research samples, or completing QOL Surveys will be reported. A few AEs were initially reported by sites but later were assessed by the Medical Monitor and determined to be report filed in error. Such AEs are not included in this report.
Arm/Group | HCT Arm | Non-HCT Arm
All-Cause Mortality (participants affected / at risk) | 125/260 | 86/124
Serious Adverse Events (participants affected / at risk) | 0/260 | 0/124
Other Adverse Events (participants affected / at risk) | 0/260 | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT02016781/Prot_SAP_ICF_000.pdf